CLINICAL TRIAL: NCT06643312
Title: Tethered Pelvic Assist Device for Recovery of Standing After Severe SCI
Brief Title: TPAD for Recovery of Standing After Severe SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Gail Forrest, Associate Director, Tim and Caroline Reynolds Center for Spinal Stimulation, Kessler Foundation
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R-1232-23
Record Dates: First submitted 2024-09-18; First posted 2024-10-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: SCI - Spinal Cord Injury
Keywords: TPAD
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: The study will include 50 participants, 20 with SCI who are able to stand independently for short periods of time (<1 hour) (Groups 1 & 3), 20 participants with SCI who are unable to stand independently (Groups 2 & 4), and 10 non-disabled individuals (Group 5). Group 1 (n=10) will be evaluated before and after receiving stand training with the TPAD. Group 2 (n=10) will be evaluated before and after receiving stand training with the TPAD. Group 3 (n=10) will be evaluated without receiving any intervention. Group 4 (n=10) will be evaluated without receiving any intervention. Groups 3 and 4, who will not receive any intervention, will undergo the Stable Standing Assessment and the Postural Perturbation Assessment only. Group 5 (n=10) will undergo assessments only. Each individual will serve as their own control, reducing the variability among individuals. Motor patterns recorded from the SCI participants will be also compared to those collected from non-disabled individuals.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (5):
- Group 1 (Other): * Individuals with SCI that can stand independently
  * Will receive TPAD training
  * Will undergo standing, posture, sitting, and stepping assessments
  * Participation in this group will last about six months
  Interventions: Device: The Tethered Pelvic Assist Device (TPAD)
- Group 2 (Other): * Individuals with SCI that cannot stand independently
  * Will receive TPAD training
  * Will undergo standing, posture, sitting, and stepping assessments
  * Participation in this group will last about 6 months
  Interventions: Device: The Tethered Pelvic Assist Device (TPAD)
- Group 3 (No Intervention): * Individuals with SCI that can stand independently
  * Will undergo standing and posture assessments
  * Participation in this group will last about 2 weeks
- Group 4 (No Intervention): * Individuals with SCI that cannot stand independently
  * Will undergo standing and posture assessments
  * Participation in this group will last about 2 weeks
- Group 5 (No Intervention): * Individuals without a SCI
  * Will undergo standing, posture, and sitting assessments
  * Participation in this group will last about 2 weeks

INTERVENTIONS:
Device: The Tethered Pelvic Assist Device (TPAD) — a light-weight cable-driven robotic stand trainer that (i) can provide assistance-as-needed by applying corrective forces on the trunk and pelvis in response to their movement outside a pre-programmed area, and (ii) can apply controlled forces on the trunk and pelvis to perturb them from their nominal configuration during standing.
  Arms: Group 1; Group 2

SUMMARY:
The purpose of this study is to investigate how standing and sitting balance control is altered after spinal cord injury (SCI) and how a new type of robotic assistive device may be used to improve muscle function. This device is called the Tethered Pelvic Assist Device, or TPAD.

The main aims are to:

1. Examine muscle activation patterns generated during different types of standing in spinal cord injured individuals using robotic assistance or self-assistance for balance

2 and 3. Examine the effectiveness of robotic-assisted stand training in the improvement of posture control during different types of standing and sitting in spinal cord injured individuals.

Participants will be placed into one of 5 groups based on a physical classification of their spinal cord injury:

Group 1:

* Individuals with SCI that can stand independently
* Will receive TPAD training
* Will undergo standing, posture, sitting, and stepping assessments
* Participation in this group will last about six months

Group 2:

* Individuals with SCI that cannot stand independently
* Will receive TPAD training
* Will undergo standing, posture, sitting, and stepping assessments
* Participation in this group will last about 6 months

Group 3:

* Individuals with SCI that can stand independently
* Will undergo standing and posture assessments
* Participation in this group will last about 2 weeks

Group 4:

* Individuals with SCI that cannot stand independently
* Will undergo standing and posture assessments
* Participation in this group will last about 2 weeks

Group 5:

* Individuals without a SCI
* Will undergo standing, posture, and sitting assessments
* Participation in this group will last about 2 weeks

DETAILED DESCRIPTION:
The investigators will be testing a device called the Tethered Pelvic Assist Device or TPAD. The TPAD provides active control and support of the trunk, pelvis, and knees during training to improve the ability to stand. Also, the TPAD can be used to safely challenge participants during standing by providing controlled "pushes" or "perturbations" that must be corrected for in order to maintain proper posture and upright balance. This could be helpful for improving muscle function after spinal cord injury.

Methodology:

The Tethered Pelvic Assist Device (TPAD) is a light-weight cable-driven robotic stand trainer that (i) can provide assistance-as-needed by applying corrective forces on the trunk and pelvis in response to their movement outside a pre-programmed area, and (ii) can apply controlled forces on the trunk and pelvis to perturb them from their nominal configuration during standing.

A total of 50 participants will be enrolled in this study; they will be broken into five groups with 10 participants in each. All participants will undergo a physical classification of their spinal cord injury to determine eligibility and which group they belong in. Group 1 will consist of individuals with SCI that can stand independently and will receive TPAD training and assessments, Group 2 will consist of individuals with SCI that cannot stand independently and will receive TPAD training and assessments, Group 3 will consist of individuals with SCI that can stand independently and will receive assessments only, Group 4 will consist of individuals with SCI that cannot stand independently and will receive assessments only, and Group 5 will consist of individuals without a SCI that will receive assessments only. Each individual will serve as their own control, to reduce variability. Motor patterns recorded from the SCI research participants will be also compared to those collected from individuals who do not have a SCI. All participants will undergo the Stable Standing Assessment and Postural Perturbation Assessment. Groups 1, 2, and 5 will additionally perform the Stable Sitting Assessment and Postural Perturbation Assessment in Sitting. Only Groups 1 and 2 will also perform the Neuromuscular Recovery Scale and attend training sessions with the TPAD system.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age at the time of enrollment;
2. stable medical condition
3. at least one year post-spinal cord injury (Groups 1-4)
4. non-progressive, traumatic SCI above T10 (Groups 1-4)
5. Injury Grade A, B, C or D (Groups 1-4)
6. ability to stand independently for short periods of time, not exceeding 1 hour (Groups 1 and 3)
7. inability to stand independently (Groups 2 and 4)

Exclusion Criteria:

1. unwillingness to wean from anti-spasticity medications;
2. untreated painful musculoskeletal dysfunction, unhealed fracture, contracture, pressure sore or urinary tract infection
3. history of bone disease unassociated with decreased bone mineral density due to spinal cord injury
4. ongoing drug abuse
5. untreated psychiatric disorders or clinical depression
6. received botox injections in lower extremities in the prior six months
7. Cardiopulmonary disease that may interfere with assessments
8. Untreated severe and persistent dysautonomia
9. Neurological injury or disease (Group 5)
10. Orthopedic injury or condition (Group 5)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Sitting Assessment | On average 4 hours to complete. Done at the beginning of the study for groups 1, 2, and 5. Repeated by groups 1 & 2 during training (up to 4 times) and at the end of the study (on average 6 months).
  Research participants will sit on a padded table and perform tasks to challenge their balance control (reaching/shifting weight in multiple directions). Assistance for sitting will be provided at the trunk by the TPAD or by the trainer. EMG and kinematic analysis will be performed on the lower extremities, trunk and upper extremities during sitting. The trunk force and position controller data from the TPAD will be also collected; these data will be synchronized with EMG and kinematic data. Muscle activation patterns will be evaluated recording EMG from different muscle groups. The TPAD/trainer will then generate controlled loss of balance during sitting. EMG onset and burst duration relative to perturbation onset, loss of balance onset and return to balance will be compared. EMG mean and integrated amplitudes from each muscle will be compared before and after training. Relationships between these parameters will also be calculated and compared with non-disabled data.
Neuromuscular Recovery Scale (NRS) | On average, 2 hours to complete. Groups 1 and 2 will complete the NRS at the beginning of the study and at the end (on average 6 months).
  Research participants will undergo a series of tasks to test the level of muscle activation and amount of assistance required during standing and stepping in a body-weight supported treadmill environment, as well as overground motor tasks. Arm, trunk/leg movement recovery and independency will be measured by the NRS using 14 motor tasks (sit, reverse sit up, sit up, sitting truck extension, overhead press, forward reach and grasp, door pull and open, can open and manipulation, sit to stand, stand, walking, stand adaptability, step retraining, and step adaptability) and combined with EMG, kinematic, and kinetic analyses on the upper and lower extremities and/or trunk. Based on the performance across categories, 4 phase scores can be assigned:1- greatest impairment relative to normal movement patterns (non-ambulatory), 2- begins to stand and weight support independently, 3- walking with varying skill levels, and 4- normal locomotor and transfer performance with adaptability.
Standing Assessment | On average 4 hours to complete. Done at the beginning of the study for all groups. Repeated by groups 1 & 2 during training (up to 4 times) and at the end of the study (on average 6 months).
  Participants will stand as long as possible and undergo a series of standing tasks. Electromyography (EMG), kinematic and kinetic analysis will be performed on the lower extremities and trunk during standing. The pelvic, trunk and knee force and position controller data from the TPAD will be collected and synchronized. Muscle activation patterns will be evaluated recording EMG from different muscle groupings. When appropriate, ground reaction forces will be measured. Blood pressure and heart rate will be measured. The TPAD will then generate controlled loss of balance during standing. Participants will regain balance with/without grasping a fixed object. Investigators will compare EMG onset and burst duration relative to perturbation onset, loss of balance onset and return to balance if applicable. EMG mean and amplitudes from each muscle will be compared before and after training. The relationship between these parameters will also be calculated and compared with non-disabled data.

CONTACTS AND LOCATIONS:
Overall Officials: Gail F Forrest, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
All Individual Participant Data (IPD) will be kept with the study research team at Kessler Foundation. IPD will be de-identified and may be shared with the device research team at Columbia University, the FDA, Kessler Foundation Institutional Review Board, the Department of Health and Human Services, and collaborators at the Kentucky Spinal Cord Injury Research Center.